CLINICAL TRIAL: NCT03279185
Title: Adolescent Master Protocol for Participants 18 Years of Age or Older - Lite (AMP Up Lite)
Brief Title: Adolescent Master Protocol for Participants 18 Years of Age or Older - Lite
Acronym: AMP Up Lite
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); NIH Office of AIDS Research (OAR) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Paige Williams, Senior Lecturer on Biostatistics, Harvard School of Public Health (HSPH)
Other Study IDs: 1P01HD103133 - PH400; PH400 (Other: PHACS Protocol Number); 1P01HD103133 (NIH)
Record Dates: First submitted 2017-08-22; First posted 2017-09-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS, perinatal HIV infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, peripheral blood mononuclear cells (PBMCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infected Cohort - closed to accrual: Perinatally HIV-infected participants at or beyond their 18th birthday at enrollment.

SUMMARY:
This is a prospective cohort study designed to define the impact of HIV infection and antiretroviral therapy (ART) on young adults with perinatal HIV infection as they transition to adulthood.

DETAILED DESCRIPTION:
This is a prospective cohort study designed to define the impact of HIV infection and antiretroviral therapy (ART) on young adults with perinatal HIV infection as they transition to adulthood.

The primary objectives of this study are:

1. To identify infectious and non-infectious complications of HIV disease and toxicities resulting from long-term ART, including disease progression, immune suppression, viral resistance, end-organ disease, and mortality.
2. To define the impact of HIV infection and ART on the long-term clinical outcomes of young adults with perinatal HIV.
3. To define the impact of perinatal HIV infection and ART on long-term mental and behavioral health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Perinatal HIV infection as documented in the medical record;
* At or beyond their 18th birthday at the time of informed consent with no upper age limit;
* Willingness to provide access to existing medical records; and
* Willingness to participate and provide legal consent

Exclusion Criteria:

* Prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Perinatally HIV-infected (PHIV+) young adults 18 years of age or older at the time of enrollment born to HIV-infected mothers.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
HIV Disease Progression | Annually for 6 years
  Factors of interest for this outcome include virologic suppression, immune impairment, immune activation, changes in ART, cumulative exposure to specific ART, viral resistance, co-infections, and host genetic polymorphisms. Data will be collected through chart abstraction.
Metabolic Anomalies | Annually for 6 years
  Data will be collected by chart review, physical assessments, and laboratory evaluations.
Sexually Transmitted Infections | Annually for 6 years
  Data collected through chart abstraction.
Reproductive Health | Annually for 6 years
  Data collected through an online surveys and chart abstraction.
Mental Health | Annually for 6 years.
  Data collected through an online survey and chart abstraction.
ART Adherence | Annually for 6 years
  Data collected through an online survey.
Risk Behaviors (Sexual and Substance Use) | Annually for 6 years
  Data collected through an online survey.
Transition to Adult Functioning | Annually for 6 years.
  Data collected through an online survey.
Hearing Dysfunction | Annually for 6 years.
  Data collected through an online survey and chart abstraction.

CONTACTS AND LOCATIONS:
Overall Officials: Paige L Williams, Principal Investigator — Harvard School of Public Health (HSPH); Katherine Tassiopoulos, DSc, MPH, Study Chair — Harvard School of Public Health (HSPH); Russell B Van Dyke, MD, Study Chair — Tulane University School of Medicine
Locations (9):
- United States (9):
  - University of Southern California, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Cook County Hospital Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New York University School of Medicine, New York, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Result] Lemon TL, Tassiopoulos K, Tsai AC, Cantos K, Escudero D, Quinn MK, Kacanek D, Berman C, Salomon L, Nichols S, Chadwick EG, Seage GR 3rd, Williams PL; Pediatric HIV/AIDS Cohort Study (PHACS). Health Insurance Coverage, Clinical Outcomes, and Health-Related Quality of Life Among Youth Born to Women Living With HIV. J Acquir Immune Defic Syndr. 2023 Jan 1;92(1):6-16. doi: 10.1097/QAI.0000000000003100. PMID 36150048
- [Result] Olivero R, Williams PL, Sawyer G, Yee LM, Patel K, Hernandez-Diaz S, Powis K, Paul M, Chadwick EG; Pediatric HIV/AIDS Cohort Study and the HOPE study. Birth outcomes following bictegravir exposure during pregnancy. AIDS. 2025 Mar 15;39(4):381-386. doi: 10.1097/QAD.0000000000004041. Epub 2024 Oct 14. PMID 39411892
- See also: Pediatric HIV/AIDS Cohort Study — http://www.phacsstudy.org